CLINICAL TRIAL: NCT01611623
Title: A Phase 1, Open-label, Dose-escalation Study of the Safety and Pharmacokinetics of SNX-5422 in Subjects With Refractory Solid Tumor Malignancies or Non-Hodgkin's Lymphoma
Brief Title: Safety and Pharmacology Study of SNX-5422 in Subjects With Refractory Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Esanex Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNX-5422-CLN1-004
Record Dates: First submitted 2012-05-25; First posted 2012-06-05 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Cancer
Keywords: Solid tumor malignancy; Hsp90
MeSH Terms: conditions — Neoplasms | interventions — SNX-5422

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SNX-5422 (Experimental): Open label administration of SNX-5422 tablets every other day for 21 days on a 28 day cycle. Dose escalation based on safety outcomes
  Interventions: Drug: SNX-5422

INTERVENTIONS:
Drug: SNX-5422 — Tablets dose every other day; dose escalation based on safety

SUMMARY:
Hsp90 is a chemical in the body that is involved in promotion of cancer. SNX-5422 is an experimental drug that blocks Hsp90. It is being evaluated for safety in patients with cancer.

DETAILED DESCRIPTION:
Correlation has been observed between Hsp90 client protein level changes and functional effects in cells in in vitro studies of SNX-5422, supporting inhibition of Hsp90 as the mechanism of action for this compound. SNX-5422 has demonstrated significant antitumor activity in mouse xenograft models of human tumors, including breast (BT474, MX-1), colon (HT29), prostate (PC3), and melanoma (A375) with multiple oral dosing regimens. This study will employ critical risk management features including the use of the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, which provides a scale for consistently grading the severity of AEs, toxicity criteria analyses for dose escalation, frequent laboratory and clinical observations, correlation of AEs with plasma concentrations of drug, monitoring of the QTc interval at appropriate time points, and a conservative dose-escalation scheme.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old histologically confirmed solid tumor malignancy refractory to available therapy or for which no therapy is available adequate organ function

Exclusion Criteria:

* CNS malignancy significant GI disease at risk for prolonged QT interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicities | First 28 day cycle
  Number of patients with dose limiting toxicities defined as Grade 3 or higher on the CTCAE version 4.03 clearly related to disease progression in each dose cohort during the first cycle of study drug administration

SECONDARY OUTCOMES:
Pharmacokinetic profiles of parent drug and metabolite | Day 1 and Day 21 first cycle
  Assessment of standard pharmacokinetic parameters including area under the plasma-concentration time curve, volume of distribution, clearance elimination half life
Number of patients with adverse events as a measure of tolerability | Day 28 of each cycle
  Frequency and severity of AEs, changes in vital signs (including self-reported pain), ECG, physical examination, and clinical laboratory parameters (clinical chemistry, hematology, and urinalysis).